CLINICAL TRIAL: NCT05355350
Title: PipEracillin/Tazobactam vs mERoPENem for Treatment of AmpC-producing Bloodstream Infections: an Extension of the Original PETERPEN Trial
Brief Title: PipEracillin/Tazobactam Versus mERoPENem for Treatment of AmpC Producing Blood Stream Infections
Acronym: SPICE-M
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No eligible patients
Sponsor: Rambam Health Care Campus (Other)
Collaborators: The Chaim Sheba Medical Center (Other); Rabin Medical Center (Other); Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, MICHAL PAUL md, Prof. Mical Paul, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0295-18-RMB
Record Dates: First submitted 2022-04-04; First posted 2022-05-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Beta Lactam Resistant Bacterial Infection; Enterobacteriaceae Infections; Bacteremia
Keywords: bacteremia; enterobacteriaceae; extended spectrum beta-lactamase; meropenem; piperacillin tazobactam
MeSH Terms: conditions — Enterobacteriaceae Infections; Bacteremia | interventions — Piperacillin, Tazobactam Drug Combination; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- piperacillin tazobactam (Experimental)
  Interventions: Drug: Piperacillin / Tazobactam Injection
- meropenem (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Piperacillin / Tazobactam Injection — 4.5 grams QID
  Arms: piperacillin tazobactam
Drug: Meropenem — 1 gram TID
  Arms: meropenem

SUMMARY:
Data regarding optimal treatment for extended-spectrum beta-lactamase (ESBL) producing Enterobacterales bloodstream infection are lacking. Observational studies show conflicting results when comparing treatment with combination beta-lactam-beta-lactamase inhibitor and carbapenems. The investigators aim to evaluate the effect of definitive treatment with meropenem vs. piperacillin-tazobactam on the outcome of patients with bacteremia due to cephalosporin-non-susceptible Enterobacteriaceae. The investigators hypothesize that piperacillin-tazobactam is non-inferior to meropenem.

DETAILED DESCRIPTION:
PeterPen-SPICE-M will expland the PeterPen trial. In PeterPen we recruit patients with bacteremia caused by 3rd generation cephalosporin-resistant E. coli or Klebsiella pneumoniae. In SPICE-M we will recruit also patients with bacteremia caused by 3rd generation cephalosporin-resistant Serratia marcescens, Providencia stuartii & rettgeri, Indole positive Proteus spp. (Proteus vulgaris), Citrobacter freundii, Enterobacter cloacae, Klebsiella aerogenes and Morganella morganii. In both trials patients will be allocated within 72 hours of blood culture taking to piperacillin-tazobactam vs. meropenem to complete at least 7 days of covering antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years)
2. New onset BSI due to Serratia marcescens, Providencia spp., Morganella morganii, Citrobacter freundii, and Enterobacter spp.in one or more blood cultures associated with evidence of infection.
3. The microorganism will have to be non-susceptible to third generation cephalosporins (ceftriaxone and ceftazidime) and susceptible to both PTZ and meropenem (see microbiological methods).
4. Both community and hospital-acquired bacteremias will be included.
5. We will permit the inclusion of bacteremias due to study pathogens with concomitant growth in blood of skin commensals considered as contaminants.

Exclusion Criteria:

1. More than 72 hr. elapsed since initial blood culture taken, regardless of the time covering antibiotics were started (up to 72 hrs.).
2. Polymicrobial bacteremia. Polymicrobial bacteremia will be defined as either growth of two or more different species of microorganisms in the same blood culture, or growth of different species in two or more separate blood cultures within the same episode.
3. Patients with prior bacteremia or infection that have not completed antimicrobial therapy for the previous infectious episode.
4. Patients with septic shock at the time of enrollment and randomization, defined as at least 2 measurements of systolic blood pressure < 90 mmHg and/or use of vasopressors (dopamine>15μg/kg/min, adrenalin>0.1μg/kg/min, noradrenalin>0.1μg/kg/min, vasopressin any dose) in the 12 hours prior to randomization. In the absence of the use of vasopressors, a systolic blood pressure <90 would need to represent a deviation for the patient's known normal blood pressure.
5. BSI due to specific infections known at the time of randomization:

   1. Endocarditis / endovascular infections
   2. Osteomyelitis (not resected)
   3. Central nervous system infections
6. Allergy to any of the study drugs confirmed by history taken by the investigator
7. Previous enrollment in this trial
8. Concurrent participation in another interventional clinical trial
9. Imminent death (researcher's assessment of expected death within 48 hrs. of recruitment) or patient in palliative care

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days from randomization
  Primary Outcome Measure
Treatment failure | 7 days from randomization]
  death OR fever > 38°C in the last 48 hours OR lack of resolution of symptoms attributed to the focus of infection OR Sequential Failure Organ Assessment (SOFA) score increasing OR positive blood cultures by the time point assessed

SECONDARY OUTCOMES:
All-cause mortality | 14 and 90 days from randomization]
  Number of deceased patients
Number of participants with treatment failure | 14 days and 30 days from randomization
  death OR fever > 38°C in the last 48 hours OR lack of resolution of symptoms attributed to the focus of infection OR Sequential Failure Organ Assessment (SOFA) score increasing OR positive blood cultures by the time point assessed
Number of participants with microbiological failure | 7 days and 14 days from randomization
  Repeat positive blood cultures with index pathogen on day 4 or later from randomization
Number of participants with recurrent positive blood cultures (relapse) | 30 days and 90 days from randomization
  recurrent positive blood cultures with the index pathogen after prior sterilization of blood cultures or after end of treatment
Number of participants with Clostridium difficile associated diarrhea | 90 days from randomization
  Diarrhea with positive Clostridium difficile toxin test
Secondary bacterial infections | 90 days from randomization
  Number of participants with a new clinically-significant infection, with or without microbiological documentation. Defined using NHSN criteria for healthcare-associated infections.
Number of participants with hospital re-admissions | 90 days from randomization
  Hospital re-admission, excluding index hospitalization
Number of participants with development of antimicrobial resistance | 90 days from randomization
  clinical isolates resistant to piperacillin/tazobactam and meropenem and any carbapenem-resistant bacteria
Carriage of carbapenemase-producing Enterobacteriaceae (CPE) and non-CPE carbapenem-resistant Enterobacteriaceae in-hospital detected by weekly rectal surveillance of carriage while in-hospital | 90 days from randomization
  New acquisition of carbapenemase-producing Enterobacteriaceae (CPE) and non-CPE carbapenem-resistant Enterobacteriaceae, detected through rectal surveillance or clinical cultures
Total in-hospital days | 30 days and 90 days from randomization
  Total of in-hospital days per participant, including all admissions
Total antibiotic days | 30 days and 90 days from randomization
  Total antibiotic days per participant within all admissions
Adverse events | 30 days
  diarrhea, liver function test abnormalities, antibiotic rash or other immediate-type allergy, acute kidney injury defined according to RIFLE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rambam Health Care Campus; Dafna Yahav, MD, Principal Investigator — Sheba Tel HaShomer Medical Campus; Alaa Atamna, MD, Principal Investigator — Rabin Medical Center, Beilinson Campus; Roni Bitterman, MD, Study Director — Rambam Health Care Campus; Noa Eliakim-Raz, MD, Study Director — Rabin Medical Center, Beilinson Campus
Locations (4):
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Sheba Tel HaShomer Medical Campus, Ramat Gan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data collected during the trial will be made available for an unlimited time period following publication of trial results. Data will be available for researchers who provide a methodologically sound proposal and contingent on both the researchers' and our ethics committee approval and the signing of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: following publication and for unlimited time
Access Criteria: proposals should be sent to the principal investigator at m_paul@rambam.health.gov.il